CLINICAL TRIAL: NCT04321733
Title: Bacteriological Study of Acute Follicular Tonsillitis in Patients Attending the ENT Outpatient Clinic of Assiut University Hospital
Brief Title: Bacteriological Study of Acute Follicular Tonsillitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Wahby Dous Hana, Principal investigator, Assiut University
Other Study IDs: Bacteriology of Tonsillitis
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Acute Follicular Tonsillitis
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — Intravenous drug intake of our drug.

SUMMARY:
The objective of the study is to answer the following questions :-

1. Is there an actual failure rate in tonsillitis treatment with amoxicillin clavulanate ? If yes,
2. What is (are) the possible reason(s) to explain it in our locality ?

DETAILED DESCRIPTION:
Tonsillitis is one of the most common diseases in the throat that occurs in the younger age group .

The predominant bacteria causing tonsillitis are group A b-haemolytic streptococci (GABHS), which are highly susceptible to the penicillin group of antibiotics.

It has been reported in the literature that the rate of penicillin failure has consistently increased from about 7% in the 1950s to almost 40% in the 2000s.

Authors propose many reasons to explain such failure rates e.g. the coexistence of oropharyngeal beta-lactamase producing bacteria .

Although there were no documented reports, it was observed that there are rising reports of failure in treatment of acute follicular tonsillitis by amoxicillin clavulanate.

ELIGIBILITY:
Inclusion criteria:

patients with acute follicular tonsillitis neither younger than five years nor older than 60 years old.

Exclusion Criteria:

1. Other causes of tonsillitis that do not cause suppuration .
2. Age below five , and above 60 years .
3. Patients who received antibiotic one week before presentation .
4. Immune compromised patients .
5. Patients with quinsy.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute follicular tonsillitis
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of the isolated organism to amoxicillin clavulanate according to culture and sensitivity test | Baseline
  throat swabs that will be taken from the tonsillar exudate, placed in sterile bottles and brought to the laboratory for Bacteriological culture of the organism and Antibiotic sensitivity tests will be done for the isolated organism(s).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brook I. Overcoming penicillin failures in the treatment of Group A streptococcal pharyngo-tonsillitis. Int J Pediatr Otorhinolaryngol. 2007 Oct;71(10):1501-8. doi: 10.1016/j.ijporl.2007.06.006. Epub 2007 Jul 17. PMID 17644191
- [Background] Casey JR, Pichichero ME. The evidence base for cephalosporin superiority over penicillin in streptococcal pharyngitis. Diagn Microbiol Infect Dis. 2007 Mar;57(3 Suppl):39S-45S. doi: 10.1016/j.diagmicrobio.2006.12.020. Epub 2007 Feb 9. PMID 17292576
- [Background] Sela S, Barzilai A. Why do we fail with penicillin in the treatment of group A streptococcus infections? Ann Med. 1999 Oct;31(5):303-7. doi: 10.3109/07853899908995895. PMID 10574501
- See also: Related Info — http://www.researchgate.net/publication/285386865_Clinical_and_Bacteriological_Study_of_Acute_Tonsillitis